CLINICAL TRIAL: NCT03221738
Title: Development of a Cognitive Behavioral Mobile App for Body Dysmorphic Disorder, and Tests of Feasibility, Acceptability, and Preliminary Efficacy
Brief Title: Smartphone-Administered App Treatment for Adults With Body Dysmorphic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Telefónica S.A. (Industry)
Responsible Party: Principal Investigator, Sabine Wilhelm, PhD, Sabine Wilhelm, Ph.D., Chief of Psychology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017P000293_A
Record Dates: First submitted 2017-07-12; First posted 2017-07-19 (Actual); Results first posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-04

CONDITIONS: Body Dysmorphic Disorders
Keywords: BDD
MeSH Terms: conditions — Body Dysmorphic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- App-Based Cognitive Behavioral Therapy (Experimental): 12-week Smartphone-delivered CBT for BDD.
  Interventions: Behavioral: App-Based Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: App-Based Cognitive Behavioral Therapy — 12-week Smartphone delivered CBT for BDD. In-person cognitive behavioral therapy (CBT) is an empirically supported treatment for BDD. The app-delivered CBT in this project includes modules such as cognitive skills (e.g., cognitive restructuring, core belief work), behavioral skills (e.g., exposure with ritual prevention), and perceptual retraining/mindfulness skills.

SUMMARY:
The investigators are developing and testing a Smartphone-based cognitive behavioral therapy (CBT) "app" for body dysmorphic disorder (BDD). The investigators hypothesize that app-based CBT for BDD will be feasible and acceptable to individuals with BDD, and will improve body image concerns and related outcomes.

DETAILED DESCRIPTION:
The primary aims of this study are to develop and test the feasibility, acceptability, and preliminary efficacy of a Smartphone-based CBT treatment for adults with BDD. This project aims to solve two healthcare problems: poor access to empirically-supportive treatment for BDD, and challenges of generalizing CBT skills outside therapy sessions. Inadequate treatment access is due to limited professionals offering this specialized treatment, economic barriers, and shame preventing sufferers from seeking in-person care. Mobile app-based CBT would solve this access gap by addressing each of these barriers. Among those who obtain CBT, practicing skills outside of therapy is critical for treatment effectiveness, as BDD symptoms occur around-the-clock and can be most impairing at home. However, BDD patients struggle to use skills without therapists' in-person support. App-based CBT that provides on-hand skills coaching addresses this treatment generalization challenge.

This study involves developing the app-based CBT for BDD treatment, and then investigating the initial feasibility, acceptability, and preliminary efficacy of the app-based treatment in an open pilot trial (N = 10), consisting of 12-weeks of active treatment plus a 6-month follow up period.

ELIGIBILITY:
Phase 1B (open pilot trial):

Inclusion Criteria:

* At least 18 years of age
* Outpatients
* Meets current diagnosis of primary DSM-5 BDD
* Has score on BDD-YBOCS of ≥ 20
* Currently living in the United States

Exclusion Criteria:

* Psychotropic medication changes within 2 months prior to enrollment
* Participants taking psychotropic medication have to have been on a stable dose for at least 2 months prior to enrollment and not change medication during study period
* Participated in CBT for BDD ever during lifetime
* Current substance dependence
* Lifetime bipolar disorder or psychosis
* Acute, active suicidal ideation
* Current severe comorbid major depression, defined by a PHQ-9 total score ≥ 20
* Personality disorder that could jeopardize treatment participation (e.g., borderline personality disorder with self-harm)
* Concurrent psychological treatment
* Do not own a supported mobile Smart phone with a data plan (currently iPhone 5S or more recent, running iOS 9 or newer)
* Intellectual disability or other cognitive impairment that would interfere with ability to engage in CBT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wilhelm, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilhelm S, Weingarden H, Greenberg JL, McCoy TH, Ladis I, Summers BJ, Matic A, Harrison O. Development and Pilot Testing of a Cognitive-Behavioral Therapy Digital Service for Body Dysmorphic Disorder. Behav Ther. 2020 Jan;51(1):15-26. doi: 10.1016/j.beth.2019.03.007. Epub 2019 Aug 7. PMID 32005333

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | App-Based Cognitive Behavioral Therapy
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | App-Based Cognitive Behavioral Therapy
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (5.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Treatment Completion Rates
Description: Number of subjects who completed the app-based treatment to assess feasibility and acceptability
Time Frame: Post treatment assessment (12 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | App-Based Cognitive Behavioral Therapy
Number analyzed (Participants) | 10
Participants | 10

2. Primary Outcome: Client Satisfaction Questionnaire (CSQ). This Measure Will be Used to Assess Change Over the Course of Treatment Twice Throughout the Study (Over Approximately 10 Months Total).
Description: The Client Satisfaction Questionnaire (CSQ) is a 25-item self-report questionnaire which assesses the satisfaction with clinical services received. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Time Frame: Post-treatment assessment (week 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | App-Based Cognitive Behavioral Therapy
Number analyzed (Participants) | 10
score on a scale | 27.90 (3.51)

3. Secondary Outcome: Yale Brown Obsessive Compulsive Scale Modified for BDD (BDD-YBOCS). This Measure Will be Used to Assess Change Over the Course of Treatment at Five Time Points Throughout the Study (Over Approximately 10 Months Total).
Description: The BDD-YBOCS is the gold-standard, semi-structured clinician-administered assessment of BDD severity. It contains 12 items ranging from 0 to 4, which are summed to generate a total score (range = 0 to 48). Higher scores indicate more severe BDD symptoms. The BDD-YBOCS will be used to assess change in BDD symptoms from baseline to endpoint.
Time Frame: Post-treatment assessment (week 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | App-Based Cognitive Behavioral Therapy
Number analyzed (Participants) | 10
score on a scale | 16.50 (3.63)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected at mid-treatment (6 weeks), post-treatment (12 weeks), 3-month and 6-month follow-up assessment time-points.
Arm/Group | App-Based Cognitive Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | App-Based Cognitive Behavioral Therapy (N=10)
Urinary tract infection (Infections and infestations) | 1 (1)
Depressive symptoms (Psychiatric disorders) | 3 (3)
Pap smear (Reproductive system and breast disorders) | 1/8 (1)
Delayed menstrual cycle (Reproductive system and breast disorders) | 1/8 (1)
Increased stress/anxiety (Psychiatric disorders) | 2 (3)
Breast lump examination (Reproductive system and breast disorders) | 1 (1)
Wisdom teeth removal (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/38/NCT03221738/Prot_SAP_000.pdf